CLINICAL TRIAL: NCT00499551
Title: A Phase I/IIa Study of the Treatment of None-infectious Anterior, Intermediate, Posterior and Panuveitis, With the Use of Dexamethasone Delivered by a Iontophoresis Device
Brief Title: A Phase I/IIa Study for the Treatment of Uveitis With Iontophoresis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The drug needed for the study is not available in Mexico anymore.
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Iontophoresis001
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Uveitis
Keywords: Anterior Uveitis; Posterior Uveitis; Intermediate Uveitis; Panuveitis; Iontophoresis; Dexamethasone
MeSH Terms: conditions — Uveitis; Uveitis, Anterior; Uveitis, Posterior; Uveitis, Intermediate; Panuveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Iontophoresis second generation Eyegate II device

SUMMARY:
The multiple properties of the corticosteroids over the inflammatory response, make them first line drugs for the treatment of several ocular inflammatory disorders of different etiologies. In order to diminish the corticosteroids severe systemic adverse effects, the local administration is preferred. Iontophoresis already has been used in a successful way for the administration of corticosteroids. Clinical or histopathological injuries due to the use of transcleral CCI have not been observed. being successful the administration of methylprednisolone by means of this system in previous studies. The objective is to evaluate the tolerance, security and effectiveness of this treatment, using a new generation device.

DETAILED DESCRIPTION:
The multiple properties of the corticosteroids on the inflammatory response, make them a first line election in the treatment of several ocular inflammatory disorders of different etiologies. Within its properties we can mention: the reestablishment of the vascular permeability, decrease of the cellular infiltrated and the exudation of fibrin, alteration of the activity of monocytes and neutrophils, decrease the proliferation of fibroblasts and endothelial cells and diminish the neovascularization post inflammation (1). For that reason, not only they diminish the inflammatory reaction, but they also diminish the formation of permanent scar, that often is responsible for the visual loss (2,3).

The most severe systemic adverse effects of the corticosteroids are: systemic hyperglicemy, the formation of gastric ulcers, avascular necrosis to of the head of the femur, suppression of the hypothalamus-pituitary adrenal axis, arterial hypertension among others (21,22). In order to diminish the severe systemic adverse effects of the corticosteroids, the local administration is preferred (4). The subconjunctival injection or topical instillation, reaches effective concentrations in the anterior chamber (5-7) whereas to reach these concentrations in the posterior segment it requires a systemic, intravitreous or periocular administration (8-11). Generally it require multiple injections, which produces patient discomfort. In addition, after periocular administration, just a small fraction of the drug penetrates the eye, whereas the rest is systemically absorbed, reason why the systemic adverse effects are not avoided.

Iontophoresis already has been successful used for the administration of corticosteroids, reaching high and lasting concentrations in both segments of the eye. (12-13). Remaining with effective concentrations up to 40 to 60 hours after the administration (23). But, Because focal chorioretinal injuries have been described, with the use of transcleral Iontophoresis, using current of high densities (14-18), this method has not gain a space in the current clinical practice. It has been previously demonstrated that the Controlled Column Iontophoresis (CCI Eyegate, Optis France SA) was as effective as the intraperitoneal administration of Dexamethasone for the treatment of the anterior and posterior uveitis induced by endotoxins (19). Through control of the electrical parameters and using safer settings, clinical or histopathological injuries due to the use of transcleral CCI have not been observed (20). The results of a pre-clinical study, in which methylprednisolone succinate by means of CCI was administered, demonstrated to be a safe method, reporting high and lasting intraocular concentrations.

In addition, a study in France was elaborated, that included 89 patients with different intraocular inflammatory diseases. Such as corneal graft rejections, previous uveitis, postoperative endophthalmitis, macular edema and inflammations of the posterior segment. For the evaluation of the security and effectiveness of the administration of methylprednisolone by means of CCI. The patients were enlisted if they required periocular or systemic treatment due to the failure of maximal topical therapy. The average of treatment with Iontophoresis was of 2,7 +/- 0,9 (1-5), with an current intensity of 1,2 to 2mA and duration of 2 to 5 minutes of each treatment.

A significant increase of conjunctival hyperemia was observed, subsequent to each CCI, which spontaneous resolved. There were no related adverse Effects. Still more, it was observed an increase of the visual acuity and decrease of the clinical inflammation in this group of patients. No of the patients loss vision and the inflammation biomarkers, taken like a whole, continued improving up to 30 days after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of, none-infectious anterior, intermediate, posterior or panuveitis, with or without associate systemic disease, like: Vogt Koyanagi Harada, Wegener Granulomatosis, Systemic erythematous Lupus, Behçet disease, etc.
* Requirement or with current topical treatment with steroids (more than every 6 hours), needs acute or chronic treatment with oral, intravenous, periocular or intravitreous corticosteroids or immunosuppressive agents for the control of the disease.
* Best Corrected Visual Acuity in the worse eye of 20/40 to 20/800 in ETDRS record.
* Patients with good mydriasis and no significant ocular opacities.
* Patients who do not plan elective surgery.

Exclusion Criteria:

* Infectious, pos-traumatic, Fuchs or self-limited uveitis. Patients with Diagnosis of glaucoma or ocular hypertension (greater than 25mmHg).
* Diagnosis or suspects ocular or central nervous system lymphoma. Patients with only one eye.
* Associated optical Neuritis of any etiology.
* Severe injuries in the eyelids or in the ocular surface that prevent the application of the electrode.
* Well-known allergy to the Dexamethasone.
* Toxoplasma scar or vitreous hemorrhage.
* Corneal injuries of herpetic origin or with suspicion of being herpetic.
* Patients with poor mydriasis, significant ocular opacities that prevents the evaluation of the posterior pole or the follow-up studies.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
to assess the tolerance, security and effectiveness in the treatment of different intraocular inflammatory disease | two years

SECONDARY OUTCOMES:
To establish the Iontophoresis utility in the drug administration in the treatment of the IID | two years
To establish the effectiveness of the CCI with Dexamethasone in the IID control | two years
To establish the security of the Dexamethasone administration with CCI in the treatment of the IID | two years
To establish the time in which the control of the ocular inflammation is succeed when using the CCI with Dexamethasone. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz-Mercado, MD, Principal Investigator — Asociación para Evitar la Ceguera en Mexico; Lourdes Arellanes, MD, Principal Investigator — Asociación para Evitar la Ceguera en Mexico; Raul Velez-Montoya, MD, Study Director — Asociación para Evitar la Ceguera en Mexico
Locations (1):
- Asociación para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Cole HP, Stallman J. Diamon DJ. High Dose Intravitreal Dexamethasone for Infections Endophthalmitis. Invest Ophthalmol Visc Sci. 1989;30:509-512.
- [Background] Schulman JA, Peyman GA. Intravitreal corticosteroids as an adjunct in the treatment of bacterial and fungal endophthalmitis. A review. Retina. 1992;12(4):336-40. doi: 10.1097/00006982-199212040-00007. PMID 1485018
- [Background] Stanbury RM, Graham EM. Systemic corticosteroid therapy--side effects and their management. Br J Ophthalmol. 1998 Jun;82(6):704-8. doi: 10.1136/bjo.82.6.704. PMID 9797677
- [Background] Leibowitz HM, Kupferman A. Periocular injection of corticosteroids: an experimental evaluation of its role in the treatment of corneal inflammation. Arch Ophthalmol. 1977 Feb;95(2):311-4. doi: 10.1001/archopht.1977.04450020112019. PMID 836214
- [Background] MCCARTNEY HJ, DRYSDALE IO, GORNALL AG, BASU PK. AN AUTORADIOGRAPHIC STUDY OF THE PENETRATION OF SUBCONJUNCTIVALLY INJECTED HYDROCORTISONE INTO THE NORMAL AND INFLAMED RABBIT EYE. Invest Ophthalmol. 1965 Jun;4:297-302. No abstract available. PMID 14326615
- [Background] Benson H. Permeability of the cornea to topically applied drugs. Arch Ophthalmol. 1974 Apr;91(4):313-27. doi: 10.1001/archopht.1974.03900060323017. No abstract available. PMID 4621283
- [Background] Barry A, Rousseau A, Babineau LM. The penetration of steroids into the rabbit's vitreous, choroid and retina following retrobulbar injection. I. Can J Ophthalmol. 1969 Oct;4(4):365-9. No abstract available. PMID 5822457
- [Background] Bodker FS, Ticho BH, Feist RM, Lam TT. Intraocular dexamethasone penetration via subconjunctival or retrobulbar injections in rabbits. Ophthalmic Surg. 1993 Jul;24(7):453-7. PMID 8351091
- [Background] Weijtens O, van der Sluijs FA, Schoemaker RC, Lentjes EG, Cohen AF, Romijn FP, van Meurs JC. Peribulbar corticosteroid injection: vitreal and serum concentrations after dexamethasone disodium phosphate injection. Am J Ophthalmol. 1997 Mar;123(3):358-63. doi: 10.1016/s0002-9394(14)70131-x. PMID 9063245
- [Background] Weijtens O, Schoemaker RC, Cohen AF, Romijn FP, Lentjes EG, van Rooij J, van Meurs JC. Dexamethasone concentration in vitreous and serum after oral administration. Am J Ophthalmol. 1998 May;125(5):673-9. doi: 10.1016/s0002-9394(98)00003-8. PMID 9625551
- [Background] Lachaud JP. [Considerations on the use of corticoids by ionization in certain ocular diseases]. Bull Soc Ophtalmol Fr. 1965 Jan;65(1):84-9. No abstract available. French. PMID 5827464
- [Background] Lam TT, Edward DP, Zhu XA, Tso MO. Transscleral iontophoresis of dexamethasone. Arch Ophthalmol. 1989 Sep;107(9):1368-71. doi: 10.1001/archopht.1989.01070020438050. PMID 2783069
- [Background] Lam TT, Fu J, Tso MO. A histopathologic study of retinal lesions inflicted by transscleral iontophoresis. Graefes Arch Clin Exp Ophthalmol. 1991;229(4):389-94. doi: 10.1007/BF00170699. PMID 1916328
- [Background] Barza M, Peckman C, Baum J. Transscleral iontophoresis of cefazolin, ticarcillin, and gentamicin in the rabbit. Ophthalmology. 1986 Jan;93(1):133-9. doi: 10.1016/s0161-6420(86)33780-1. PMID 3951811
- [Background] Barza M, Peckman C, Baum J. Transscleral iontophoresis of gentamicin in monkeys. Invest Ophthalmol Vis Sci. 1987 Jun;28(6):1033-6. PMID 3583629